CLINICAL TRIAL: NCT05168085
Title: Randomised Controlled Trial to Test and Build Evidence Base for Providing Eggs as an Early Complementary Food to Promote Child Growth: Eggcel-growth Study
Brief Title: Efficacy of Providing Eggs as an Early Complementary Food to Promote Child Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North-West University, South Africa (Other)
Responsible Party: Principal Investigator, Marius Smuts, Professor, North-West University, South Africa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eggcel-growth
Record Dates: First submitted 2020-02-13; First posted 2021-12-23 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Linear Growth
MeSH Terms: interventions — Eggs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): One chicken egg per day
  Interventions: Dietary Supplement: Eggs
- Control group (No Intervention): True control

INTERVENTIONS:
Dietary Supplement: Eggs — Providing 1 egg per day fo 6 months to infants
  Arms: Intervention group

SUMMARY:
This study will investigate the efficacy of providing one chicken egg per day for a period of 6 months, beginning at the age of 6 to <9 months on the growth, motor development, micronutrient, and morbidity status of infants from a low socioeconomic community in South Africa.

DETAILED DESCRIPTION:
The nutritional benefit of eggs, in particular chicken eggs is well documented. However, there is paucity of evidence regarding including eggs, in particular chicken eggs during the early complementary feeding phase to enhance child growth and development. Thus, this study seeks to determine and to provide evidence on the effectiveness of including chicken eggs as an early complementary food to enhance early child growth and development. This randomised controlled trial will contribute towards building a strong evidence for the promotion and use of eggs as a healthy and nutritious early complementary food, and can be used to inform future programming regarding infant and young child feeding in low- and middle-income countries.

This is a randomised controlled trial with a parallel design (2 groups). Five hundred infants aged 6 to <9 months will be included. Infants with egg allergy or sensitization will be excluded. Data will be collected in three months' interval for six months. At baseline, body measurements of mother and infant will be taken; infant's dietary intake using 24-hour recall methods; breastfeeding and complementary feeding practices; infant and maternal allergy and maternal depression with structured questionnaires. Morbidity symptoms and compliance will be recorded daily and followed up weekly. Developmental milestones will be assessed weekly using Pictorial Gross Motor Milestone Chart. Household food security will be assessed. Capillary blood will be collected by means of finger and/or heal prick. This will be a community driven project. Data will be analysed according to intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Resident in the study municipality; Infants aged 6 to <9 months

Exclusion Criteria:

* Severe obvious congenital abnormalities such as cleft lip and spina bifida; Severe anaemia (haemoglobin <70 g/L); Severe acute malnutrition (weight-for-length z-score < -3); Plans to move out of the study area in the next nine months; Known allergies/intolerances to eggs; Infants receiving special nutritional supplements as part of feeding programmes; Not been born as a singleton; Mother/legal guardian below 18 years old at the start of the study

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 655 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Linear growth by measuring length | 6 months
  Efficacy of providing one chicken egg per day on linear growth and stunting prevalence compare to a control

SECONDARY OUTCOMES:
Motor development using Pictorial Gross Motor Milestone Chart | 6 months
  Effects of consuming one chicken egg per day on motor development compare to a control
Biomarkers of anaemia, iron, vitamin A and essential fatty acids | 6 months
  Effects of consuming one chicken egg per day on biochemical biomarkers compare to a control
Morbidity status | 6 months
  Effects of consuming one chicken egg per day on morbidity symptoms compare to a control

CONTACTS AND LOCATIONS:
Overall Officials: Marius Smuts, PhD, Principal Investigator — Director
Locations (1):
- Jouberton area in the Matlosana sub-district, Klerksdorp, North West, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakiranda R, Malan L, Ricci H, Kruger HS, Nienaber A, Visser M, Ricci C, Faber M, Smuts CM. Daily Complementary Feeding With Eggs Improves Fibroblast Growth Factor 21 in Infants. Matern Child Nutr. 2025 Apr;21(2):e13782. doi: 10.1111/mcn.13782. Epub 2024 Dec 9. PMID 39648796
- [Derived] Ricci H, Faber M, Ricci C, Kruger HS, Malan L, Nakiranda R, Visser M, Smuts CM. Effects of egg as an early complementary food on growth of 6- to 9-month-old infants: a randomised controlled trial. Public Health Nutr. 2023 Nov 29;27(1):e1. doi: 10.1017/S1368980023002604. PMID 38018158